CLINICAL TRIAL: NCT00261170
Title: Bupropion for Hospital-Based Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Joan Kaiser, Contracts & Grants, University of California Office of the President Special Research Programs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12RT-0148; 12RT-0148
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Smoking
Keywords: smoking
MeSH Terms: conditions — Smoking | interventions — Bupropion; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): bupropion and behavioral counseling
  Interventions: Drug: bupropion
- 2 (Placebo Comparator): placebo medication
  Interventions: Other: placebo

INTERVENTIONS:
Drug: bupropion — 150 mg daily for the first 3 days, then 150 mg twice daily for 7 weeks
  Other Names: Zyban
  Arms: 1
Other: placebo — 1 pill daily for the first 3 days, then one pill twice daily for 7 weeks
  Other Names: sugar pill
  Arms: 2

SUMMARY:
This is a randomized blinded trial of whether hospitalized smokers who are randomly assigned to receive bupropion, an antidepressant, and cognitive-behavioral counseling, are more likely to have quit smoking at the end of treatment and at 6 months compared with smokers randomly assigned to receive placebo and cognitive-behavioral counseling. Because depression is more prevalent among smokers and because smokers who are prone to depression may become depressed when they quit, the hypothesis is that the proportion of quitters who receive the active drug/antidepressant will be greater than the proportion of quitters who receive the placebo drug at 6 months.

DETAILED DESCRIPTION:
Two hundred and seventy patients will be enrolled;approximately 135 will be randomized to each study arm over the course of 24 months. Patients will be considered smokers if they have used tobacco products during the week prior to admission and if they have smoked> or = 5 cigarettes /day during the previous year.Smokers will be identified by review of admissions and given a flyer to invite them to join the study. Interested smokers will be screened and asked to fill out a Beck Depression Inventory. Patients with very high Beck Depression Inventory Scores, i.e. > or = 30, will not be enrolled because such individuals may require other treatment. Each patient's physician will be contacted to verify his/her eligibility for the study. Once eligibility has been ascertained, a research associate will visit the patient to obtain informed consent and to enroll them in the study. Study questionnaires and a Fagerstrom test for Nicotine Dependence will be completed and reviewed by a research associate for completeness at the time of enrollment. The associate will put in the prescription for the study drug and request the order for dispensing of the drug. The research pharmacist will randomize the patient to Study Arm 1 or Study Arm 2.

Subjects randomized to Study Arm 1 will receive a standard 7-week course of sustained release bupropion (150 mg/day for the first 3 days, then 150mg BID), a self-help booklet, counseling on smoking cessation strategies, and follow-up phone counseling during the first 3 months after randomization. Study Arm 2 participants will receive the same intervention as Study Arm 1, but will receive placebo instead of active bupropion therapy. Both study groups will complete study questionnaires regarding their medical and smoking history and will be followed one week after their hospital discharge to record their blood pressure and to monitor possible side effects.

Since quit rates tend to decline over time, relapse prevention approaches will be included in both study arms. Marlatt's theory of relapse, an extension of Bandura's social learning model, will be used to augment the quitter's perception of self-efficacy. Participants will be trained to resist and cope with the temptations and stresses likely to be encountered after discharge from the hospital. Behavioral self-management techniques to counter known relapse-triggers such as stress, the presence of other smokers, alcohol use and depression will be discussed during follow-up counseling calls.

We will measure saliva cotinine in all participants who give a history of smoking abstinence at the end of treatment and at 6 months. Cotinine levels of > or + 15 ng/mL will be considered evidence of current tobacco use. Participants who are self-reported quitters, but have failed to provide a saliva sample will be considered as smokers unless verification from a spouse or significant other can be obtained. Participants who have died will be analyzed as smokers or quitters based on prior self-report, information in medical records, or interviews with next-of-kin. Others will be censored (i.e. excluded from the analysis). All cotinine samples will be assayed at the University of California, San Francisco,laboratory of Dr. Neal Benowitz.

ELIGIBILITY:
Inclusion Criteria:

* currently smoking - use of tobacco products during the week prior to hospital admission and having smoked at least 5 cigarettes /day during the past year
* eligibility to receive medical care in a VA hospital
* hospitalization for at least 48 hours to provide sufficient time to identify, screen, enroll and counsel participants
* willingness to participate and give informed consent

Exclusion Criteria:

* hospitalization for acute CHD syndromes
* contraindications to the use of bupropion
* family history of seizure disorder, history of severe head trauma, predisposition to seizures
* unstable psychiatric disorder
* pregnancy, lactation
* current alcohol (defined as greater than 3 drinks/day) or drug abuse (defined as current/within last 3 months use of narcotics, heroin, cocaine, amphetamines)
* current untreated depression (BDI score > or = 30)
* terminal illness
* inability to be contacted by phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2003-07; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Smoking status at 6 months after enrollment | 6 months

SECONDARY OUTCOMES:
smoking status at end of treatment | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Simon, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961